CLINICAL TRIAL: NCT04576286
Title: Holmium Versus Bipolar en Bloc Transurethral Resection of Urothelium Tumor of the Urinary Bladder: A Randomized Controlled Trial
Brief Title: Holmium Versus Bipolar en Bloc Transurethral Resection of Urothelium Tumor of the Urinary Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R32/2020
Record Dates: First submitted 2020-09-16; First posted 2020-10-06 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Urinary Bladder Neoplasm
Keywords: urinary bladder tumors; en bloc resection; holmium laser; bipolar; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent, patients will be randomized with a 1:1 ratio using sealed envelopes that will be prepared by the department's ethical committee into 2 groups, group 1 represent the Holmium en bloc resection procedure while group 2 represents bipolar en bloc resection. Patients will be blinded to the type of intervention as well as the data collector and the statistician.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the type of intervention as well as the data collector and the statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium en bloc resection (Experimental): Holmium en bloc resection procedure will be done under either general or spinal anesthesia, using a Holmium laser device (Cyber Ho, Quanta device, Milano, Italy). We will use a 30-40-watt power, 1-2 joules and 20-30 MHz frequency
  Interventions: Procedure: Holmium versus Bipolar en bloc transurethral resection
- bipolar en bloc resection (Active Comparator): bipolar en bloc tumor resection of urinary bladder tumors
  Interventions: Procedure: Holmium versus Bipolar en bloc transurethral resection

INTERVENTIONS:
Procedure: Holmium versus Bipolar en bloc transurethral resection — After obtaining informed consent, patients will be randomized with a 1:1 ratio using sealed envelopes that will be prepared by the department's ethical committee into 2 groups, group 1 represent the Holmium en bloc resection procedure while group 2 represents bipolar en bloc resection. Patients will be blinded to the type of intervention as well as the data collector and the statistician.
  Intervention: all procedures will be done by an expert surgeon who performed over 50 cases of en bloc urinary bladder tumor resection with each energy source. In group A, Holmium en bloc resection procedure will be done under either general or spinal anesthesia, using a Holmium laser device (Cyber Ho, Quanta device, Milano, Italy). We will use a 30-40-watt power, 1-2 joules and 20-30 MHz frequency for Group A and bipolar en bloc resection for Group B. A 550 nm flexible laser fiber will be used in group A and a bipolar resection loop for group B.

SUMMARY:
En bloc resection of bladder tumors (ERBT) may improve staging quality and perioperative morbidity and influence tumour recurrence

DETAILED DESCRIPTION:
Modern laser technology has led to new alternatives to conventional TURBT (cTURBT). The advocates of ERBT have three goals: to improve resection quality, lower perioperative complication rates, and decrease recurrence rates at resection sites. The present study is the first to compare the results of laser and electric en bloc resection of bladder cancer with respect to the aforementioned goals.

the investigators aim to compare the clinical outcome in the form of safety and efficacy between Holmium and bipolar transurethral en bloc resection of urinary bladder tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes presented with urinary bladder tumor aiming for complete resection as diagnosed by Ultrasound with or without CT prior histopathological assessment.

Exclusion Criteria:

* Patients with signs of extravesical tumor extension where complete resection will not beneficial or unable to proceed to complete resection due to huge tumor burden either huge single tumor more than 5 cm or multiple tumors that are not candidate for complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
number of participant with Conversion to the TURBT | intraoperative finding
  conversion from the enbloc way of resection to the standard trans-urethral resection of bladder tumors

SECONDARY OUTCOMES:
Operative time | intraoperative finding
  calculation of operative time in minutes
Presence of detrusor muscle in resected sample | one day after surgery during pathological evaluation
  presence of muscle layer in the pathological specimen (Yes/No)
Resected specimen's edge | one day after surgery during pathological evaluation
  tumor free margin (Yes/No)
intraoperative complication: bladder perforation | intraoperative
  (Yes/No) bladder perforation
Incidence of obturator reflex | intraoperative
  (Yes/No) energy induced obturator reflex
hematuria | postoperative complication up to 2 weeks
  (Yes/No)
Post-operative catheterization time in hours | postoperative complication up to 2 weeks
  time till catheter removal in days
Postoperative irrigation time in hours | postoperative in hours maximum 1 day
  hours for the need of postoperative irrigation
Recurrence rate of tumors according to time interval | 1 year
  recurrence of tumor in the follow up cystoscopy
Recurrence rate of tumors according to tumor location | 1 year
  recurrence of tumor in the follow up cystoscopy in the same site or in different site

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04576286/Prot_000.pdf